CLINICAL TRIAL: NCT06871137
Title: Healthier Wealthier Families in East London (HWFinEL): Evaluating and Extending Health and Wellbeing Benefits of Universal Co-located Money Advice for Parents of Newborns
Brief Title: Healthier Wealthier Families In East London: HWFinEL
Acronym: HWFinEL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CCTU/2023/464; NIHR158551 (Other Grant/Funding Number: National Institute for Health and Care Research (NIHR))
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Mental Health; Financial Wellbeing
Keywords: Tower Hamlets; Welfare Benefits Advice; Financial Wellbeing; Financial Support for Parents; Money Advice for Parents; Benefits and Entitlements; Mental Health and Wellbeing
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: HWFinEL is a randomised controlled trial with appropriately blinded statisticians and health economists during the conduct of the study. All analyses will be conducted by suitably qualified and experienced statisticians according to a detailed prespecified statistical analysis plans (SAP).
  Participants will be randomised, after completion of their baseline questionnaire, in a 1:1 ratio to the intervention group or the control group and will be unblinded to their group allocation. Participants who are randomised to the intervention group will be contacted by telephone (by a UCL Researcher) and invited to attend a Welfare Benefits Advice (WBA) appointment within 3 months of randomisation.
  Participants who are randomised to the control group will be emailed or posted a card to their address detailing existing 'service as usual' WBA services.
  All participants will be required to complete a baseline questionnaire and a 6-month follow-up questionnaire upon study completion.
Who Masked: Outcomes Assessor
Masking Description: As above, analysing statisticians and health economists will be masked to treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1. Intervention (Other): Participants who are randomised to receive the intervention (Welfare Benefits Advice (WBA)) will be contacted by a UCL researcher and invited to attend a Welfare Benefits Advice appointment within 3 months of randomisation, to coincide with their new-born's 6-8 week health check.
  Interventions: Other: Welfare Benefits Advice (WBA)
- Arm 2. Control (Other): Participants who are randomised to the control group will be emailed or posted a card detailing the London Borough of Tower Hamlet's existing 'service as usual' Welfare Benefits Advice services, which reproduces what is available on their website.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Welfare Benefits Advice (WBA) — Appointment offered to receive financial advice from a Welfare Benefits Advisor (WBA) co-located with routine 6-8 week newborn health checks
  Arms: Arm 1. Intervention
Other: Usual care — No intervention, existing London Borough of Tower Hamlets 'service as usual'
  Arms: Arm 2. Control

SUMMARY:
The financial condition children live in when they are young can affect their health, not only in their childhood but also throughout their lives. The cost-of-living crisis means many families are 'going without' the basics. Many people do not claim all the benefits they are entitled to, or know how to solve money problems because they find it difficult to access advice. Parents with a new-born baby are especially likely to need financial support.

Research shows that after getting money advice services linked up with routine health services, family income can improve. The investigators don't yet know if linking up money advice with routine health appointments improves parents' health and wellbeing as well as their household income. The investigators don't know whether making these services easy to access through linking them up has long term implications for children's health and wellbeing. Finally, at the moment the investigators don't know how best health and money advice services can be organised to help mothers or fathers who are in difficulty such as those who are homeless or have recently arrived in England.

The goal of this trial is to improve low-income families' living conditions and ensure that all children have the best start in life. The investigators hypothesise a co-located approach will serve as a vital step toward a more integrated approach to health and social welfare, ultimately benefitting families in need. The investigators will be comparing one group of participants who will receive welfare benefits advice from a welfare benefits advisor (WBA) that is co-located with routine 6-8 week newborn health check appointments in a Children and Families Centre (CFC). The other group will receive standard care and be given information on where they can access welfare benefits advice.

DETAILED DESCRIPTION:
The trial is evaluating the impact of co-located welfare benefits advice with Health Visiting appointments and the investigators will triangulate findings from the following aspects:

* A randomised controlled trial assessing the impact of money advice services on parental mental health.
* A process evaluation to assess how the intervention is implemented and how it impacts on users.
* An economic evaluation to assess the cost-benefit of the intervention.

The overall project includes four integrated work packages (WP):

* WP1 will include a process evaluation, explore service uptake and qualitative experiences of the service.
* Findings from WP1 will be used in modelling to estimate the long-term multi-sector costs and benefits of the service (WP2).
* The investigators will use qualitative methods to co-design a draft toolkit based on the experiences and participation of a marginalised group of mothers to inform service development (WP3).
* Evidence arising from WPs1-3 will be actively disseminated locally, regionally and nationally, across a range of stakeholders, and via international networks, to maximise impact (WP4).

This is a randomised controlled trial whereby participants will be randomised in a 1:1 ratio to either the intervention group (welfare benefits advice (WBA) appointment) or the control group (existing service as usual).

The intervention will be WBA co-located with routine health appointments and delivered in Children and Families Centres (CFCs) in The London Borough (District) of Tower Hamlets. Over 98% of new babies are enrolled in the health visiting service. Co-located Welfare Benefits Advice with health appointments is an example of a Health Justice Partnership found to be an effective tool in addressing health equity.

The project will run over a period of 36 months. The target sample size is 1153 participants. The investigators will recruit over 16 months, with a 6 month internal pilot. Participants will be followed up for 6 months from the baseline time point (though could be in the trial for up to 9 months if they consent to take part in an interview (only a sub-group of participants)).

ELIGIBILITY:
Inclusion Criteria:

* Mothers or fathers aged 16 years or over.*
* Mothers or fathers with a live baby/babies less than three months old who are registered with the health visitor service in LBTH, at the point of consent, who respond Yes to a screening question asking if they wish to receive advice about money.**
* Able to provide informed consent.
* Able and willing to complete questionnaires.

Please note:

*Only one parent will be recruited. If one parent is under the age of 16, they will not be eligible.

**If the participant has multiple children, at least one child must be <3 months old.

Exclusion Criteria:

Mothers or fathers with:

* Any known safeguarding concern.
* Maternal or paternal diagnosis of learning difficulty that affects the capacity to consent.
* A baby/babies who have significant medical complications (e.g., inpatient on a neonatal unit).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1153 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Difference in depression scores at 6 months | Six months from baseline
  Difference in depression (Patient Health Questionnaire Depression Scale-8 (PHQ-8)) scores at 6 months' follow-up in the intervention arm compared with the control arm accounting for baseline values and adjusted for stratification variables (if any). The outcome will be examined to ensure that it meets the assumptions for regression analyses and transformed, if necessary, to an appropriate scale so that the resultant distribution approaches normality.
  The PHQ-8 is an 8-item instrument with a 4-item scale. Each item asks the individual to measure their depression symptoms over the past two weeks. Response options include 0 = not at all, to 3 = nearly every day. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Financial gain at 6 months | Six months from baseline
  Difference in household financial income at 6 months' follow-up in the intervention arm compared with the control arm accounting for baseline values and for stratification values (if any). The outcomes will be examined to ensure that it meets the assumptions for regression analyses and transformed, if necessary, to an appropriate scale so that the resultant distribution approached approaches normality.
Anxiety scores at 6 months | Six months from baseline
  Difference in the General Anxiety Disorder-7 (GAD-7) scores at 6 months follow-up in the intervention arm compared with the control arm accounting for baseline values. The GAD-7 measure, is a 7-item instrument with a 4-item scale. Each item asks the individual to measure their anxiety symptoms over the past two weeks. Response options include 0 = not at all, to 3 = nearly every day. Higher scores mean a worse outcome.
Quality of Life at 6 months | Six months from baseline
  Parental wellbeing: Difference in the Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) scores at 6 months follow-up in the intervention arm compared with the control arm accounting for baseline values. The SWEMWBS is a 7-item scale with five response options. Each item asks the individual to measure their mental wellbeing over the past two weeks. Response options include 1 = none of the time, to 5 = all of the time. Higher scores mean a worse outcome.
Quality of life (economic evaluation) at 6 months | Six months from baseline
  Difference in EuroQol-5 Dimension 5-level (EQ-5D-5L) scores at 6 months follow-up in the intervention arm compared with the control arm accounting for baseline values. It comprises of 5 dimensions of health (mobility, self-care, usual activities, pain or discomfort, and anxiety or depression) with 5 levels of severity in each dimension (no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems). Higher scores mean a worse outcome.

IPD SHARING:
Plan to Share IPD: Undecided
The sharing of individual participant data is not planned outside of the direct research team (or healthcare professionals who will be seeing the participant).